CLINICAL TRIAL: NCT07253753
Title: Phase 1 Evaluation of Novel Imaging Diagnostic Agent NeuCaVis in Healthy Volunteers
Brief Title: A Study to Evaluate Safety and Dosimetry of [18F]4-FDF, a New PET Imaging Agent for Inflammation
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yellowbird Diagnostics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: YB-NCV-001
Record Dates: First submitted 2025-11-14; First posted 2025-11-28 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active (Experimental): NeuCaVis
  Interventions: Drug: NeuCaVis

INTERVENTIONS:
Drug: NeuCaVis — PET radiotracer

SUMMARY:
A standard imaging test used to look for disease in the body is a positron emission tomography (PET) scan. These scans use a small amount of a radioactive substance, called a radiotracer. The most commonly used radiotracer is FDG, which shows us how the body uses glucose (a type of sugar). However, because the brain and heart naturally use a lot of glucose, the images can have background 'noise' making it harder for doctors to see signs of disease in these organs.

NeuCaVis is a new type of radiotracer that is being investigated in this study. It works by showing us how the body uses different kind of sugar, fructose. Outside of the digestive system, fructose is not normally used by healthy tissues. It is only used for energy when inflammation is present.

The purpose of this study is to evaluate the safety, tolerability and how NeuCaVis is distributed in normal tissue throughout the body. This is the first time this is being tested in people.

Participants will undergo a series of PET/CT scans following an intravenous injection of NeuCaVis. The first will be 90 minutes, then a 25 minute break, followed by a 10 minute scan, a 105 minute break, then a final 10 minute scan. A follow up phone call will occur 1-3 days later. In the optional sub-set study, participants will return to the clinic approximately 1-2 weeks after the first scan. The additional PET scan is already used in medical care and involves administration of an approved PET radiotracer, [18F]FDG. Researchers would compare this scan to the study PET scan with NeuCaVis. For this standard of care scan, it would be necessary to fast (not to eat or drink anything, except water) for at least 12 hours prior to receiving the FDG radiotracer injection.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ages 18-55 years inclusively at time of consent
2. Body Mass Index (BMI) of 18 to 30 kg/m2, inclusively
3. Capable of providing informed consent
4. Able to speak and read in English or French
5. Able to comply with all study procedures (including fasting for 12 hours, lying still in a supine position for about 90 minutes)

Exclusion Criteria:

1. Known hypersensitivity NeuCaVis or its excipients
2. Blood glucose level higher than 200mg/dl at screening
3. Active viral infection at screening
4. Currently taking anti-inflammatory medications (e.g. ASA, NSAIDs, corticosteroids, immunomodulating agents, colchicine)
5. Any anatomical heart abnormality, or cardiovascular condition including acute cardiac condition, suspicion of cardiac inflammation, and/or coronary artery disease, that may confound the analysis of the data based on the investigator's clinical opinion.
6. Recent (in the past 6 months) history of head trauma
7. Abnormal and clinically significant results on the physical examination, vital signs, or laboratory tests at screening.
8. Clinically significant neurologic, neurodevelopmental, cardiovascular, renal, hepatic, hematological, gastrointestinal, pulmonary, or metabolic-endocrine disorder
9. Female participants who are pregnant, planning to become pregnant during the study or breastfeeding
10. If of childbearing potential, unwilling or unable to use of a highly effective method of contraception as outlined in the protocol for the duration of the study.
11. Any contraindication to PET or CT imaging.
12. Actively participating in other interventional clinical trial(s).
13. Unwilling to comply with study procedures, medication restrictions or attend all study visits
14. Any other condition that, in the opinion of the investigator, could create a hazard to the participant's safety, endanger the study procedures, or interfere with the interpretation of study results.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events (TEAEs) and treatment emergent serious adverse events (TESAEs) | Adverse events are collected on each day participants undergo PET scanning (Day 1 and optional sub-study Day 8-15) and at safety follow-up visits two days post scanning.
  Categorized by type, severity and relationship

SECONDARY OUTCOMES:
Radiotracer uptake measured in major organs | Day 1
  Measured by SUV and mean uptake time for radiotracer. Visual analysis for any non-physiological radiotracer uptake.
Whole blood and plasma radioactivity counts | Day 1
  Measured at 0.5 to 250 min post-injection. Time-activity curves (TACs) for major organs.
Overall visual grading score | Day 1
  Measured by present or not present
Qualitative scoring scale | Day 1
  Measured by none (0), minimal (1), mild (2), moderate (3), severe (4) for LV myocardium
Image quality | Day 1
  Measured by non-diagnostic (0), poor (1), fair (2), good (3), excellent (4)
Cardiac and brain uptake | Day 1
  Measured by none (0), minimal (1), mild (2), moderate (3), extreme (4)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Chow, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No